CLINICAL TRIAL: NCT06040554
Title: The Effect Of A Resistance Exercise Program On Balance Of Elderly People: A Pilot Trial
Brief Title: The Effect Of A Resistance Exercise Program On Balance Of Elderly People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of West Attica (Other)
Responsible Party: Principal Investigator, Kontonikas Konstantinos, Principal Investigator, University of West Attica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UWestAttica
Record Dates: First submitted 2023-09-06; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Aging Well; Aging
Keywords: aging; elderly; strength; balance; elastic band

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Program (Experimental): Participants will participate in a group resistance exercise program for 8 weeks, using elastic bands.
  Interventions: Other: Elastic Band Resistance Exercises
- Unchanged Activities of Daily Living (No Intervention): Participants will be asked not to change their activities of daily living for the duration of the research.

INTERVENTIONS:
Other: Elastic Band Resistance Exercises — 8 Warm-Up Exercises followed by 10 Elastic Band Exercises followed by 8 Post-Workout Exercises.
  Arms: Exercise Program

SUMMARY:
The purpose of the present study is to investigate the effectiveness of a resistance exercise program consisting of elastic band exercises to balance, strength and quality of life of community-dwelling elders. The hypothesis of the study is that the people training with elastic bands will show benefits on the aforementioned areas.

DETAILED DESCRIPTION:
The elderly are, according to research, prone to an accelerated rate of loss of balance, particularly after the age of 60. This loss of balance could translate to injurious falls which could lead to trauma, fear of falling or even hospitalization. It has been shown in multiple studies that strength training can provide health benefits to the general population improving strength, balance, postural control, bone health and quality of life.

Elastic band exercises could be applied to a number of different settings due to the comparably low cost of equipment and due to the easiness of handling the equipment. In previous studies, elastic band exercise programs, varied in design, have been shown to provide multiple benefits to elderly people. In this study, it is proposed that in a Community Center for Elderly People, which are widely established in Greece, a group of eligible community dwelling elderly could exercise under supervision using elastic bands in a group setting.

The recruitment will take place in a Community Center for Elders. A group of people aged over 65, able and cleared to participate in strength training will participate. Information sheet and consent form will be provided to all participants. A pilot randomized intervention study is designed to assess the efficacy of elastic band resistance training as means to improve balance, strength and quality of life where the sample will be randomized to one of two following study groups:

1. exercise program group (intervention group)
2. no change of activities of daily living (control group)

Assessment will be obtained in two-time periods: prior to the program and after the program.

The exercise program will take place twice-weekly for eight weeks.

Participants will be assessed using Berg Balance Scale, Gait Speed, Timed Up and Go, 30 Seconds Chair Stand Test, Handgrip Strength, Knee Extensors and Flexors Strength, Fall Efficacy Scale.

ELIGIBILITY:
Inclusion Criteria:

* Over 65 years old
* Able to consent to participation
* Able to stand without assistive devices
* Able to participate in strength training
* Able to perform activities of Daily Living independently
* Cognitively and psychologically able to participate in a group setting

Exclusion Criteria:

* Systematically exercised for up to 6 months prior to start of study
* Neurological disorders or inability to stand
* Recent surgery or contraindications to exercise
* Arthroplasty or Prosthetic Limbs
* Vision or Hearing problems hindering participation in group
* Medication or Disorders contraindicating exercise or standing
* Hypotension or Orthostatic Hypotension
* Malignancy or Recent Treatment for Malignancy

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-20 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | At baseline and after the end of the 8th week of the training program, at week number 9
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. It does not include the assessment of gait.

SECONDARY OUTCOMES:
Gait Speed 4 Meters | At baseline and after the end of the 8th week of the training program, at week number 9
  The speed with which a patient walks for 4 meters. Gait speed is a metric that is extremely valuable for practitioners when examining aspects of functional mobility in their patients. Additionally, given its ability to be influenced by multiple body systems (i.e. central nervous system, musculoskeletal system), gait speed is often used as a predictor of overall health and function, especially in older adults.
Timed Up and Go | At baseline and after the end of the 8th week of the training program, at week number 9
  The patient is asked to stand from a sitting position, walk for three meters, turn around and return to seat. The purpose of this is to determine fall risk and measure the progress of balance, sit to stand and walking. It is a simple screening test that is a sensitive and specific measure of probability for falls among older adults.
30 Seconds Chair Stand Test | At baseline and after the end of the 8th week of the training program, at week number 9
  Patient is asked to alternate between sitting and standing for 30 seconds. The 30 second chair stand test is for testing leg strength and endurance in older adults.
Handgrip Strength | Prior to the 1st week of the training program, After the end of the 8th week of the training program
  Grip Strength is measured by use of a Grip Dynamometer. Grip strength is a measure of muscular strength or the maximum force/tension generated by one's forearm muscles. It can be used as a screening tool for the measurement of upper body strength and overall strength.
Lower Limb Strength (Flexors - Extensors of Knee) | At baseline and after the end of the 8th week of the training program, at week number 9
  Muscle Strength will be measured by use of Dynamometer. An assessment of muscle strength is typically performed as part of a patient's objective assessment and is an important component of the physical exam that can reveal information about neurologic deficits. It is used to evaluate weakness and can be effective in differentiating true weakness from imbalance or poor endurance.
Fall Efficacy Scale International (FES-I) | At baseline and after the end of the 8th week of the training program, at week number 9
  The Falls Efficacy Scale International (FES-I) is a measure of "fear of falling" or "concerns about falling", developed as a part of the Prevention of Falls Network Europe (ProFaNE) project from 2003 to 2006 by Todd et al. It is a 16 item questionnaire, useful to the researchers and clinicians interested in fear of falling, with a score ranging from minimum 16 (no concern about falling) to maximum 64 (severe concern about falling). The FES-I is intended to be used in adult population to measure the level of concern about falling during social and physical activities inside and outside the home whether or not the person actually does the activity.

CONTACTS AND LOCATIONS:
Overall Officials: K Kontonikas, Principal Investigator — University West Attica
Locations (1):
- Elderly Community Center, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No